CLINICAL TRIAL: NCT01983605
Title: Left Atrial Appendage Exclusion Study II
Brief Title: Left Atrial Appendage Exclusion Study
Acronym: PLACE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RS-001 V3.0_120709
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2016-10

CONDITIONS: Atrial Appendage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): LAA exclusion with the LARIAT Suture Delivery Device
  Interventions: Device: LARIAT Suture Delivery Device

INTERVENTIONS:
Device: LARIAT Suture Delivery Device — LAA exclusion procedure

SUMMARY:
Evaluate the safety and effectiveness of the LARIAT Suture Delivery device in excluding the left atrial appendage in 100 patients.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of the SentreHEART suture delivery system for the exclusion of the left atrial appendage in up to 100 treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age
2. Subject has atrial fibrillation (paroxysmal or persistent)
3. Subject is poor candidate for Warfarin (contraindicated, labile INR, non-compliant)
4. Subject is willing and able to provide written informed consent
5. Subject has a life expectancy of at least 1 year
6. Subject is willing and able to return for scheduled follow up visits

Exclusion Criteria:

1. Previous cardiac surgery
2. Thrombus in the left atrial appendage or left atrium
3. NYHA Class IV heart failure symptoms
4. Need for emergent cardiac surgery (i.e. cardiogenic shock)
5. LAA is not appropriate for exclusion based upon intraoperative evaluations
6. Current diagnosis of active systemic infection
7. Renal failure requiring dialysis or hepatic failure
8. A known drug and/or alcohol addiction
9. Mental impairment or other conditions, which may not allow subject to understand the nature, significance and scope of the study
10. Pregnancy or desire to get pregnant within 12 months of the study treatment
11. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
12. Patients who have been treated with thoracic radiation
13. Patients in current chemotherapy
14. Patients on long-term treatment with steroids not including intermittent use of inhaled steroids for respiratory diseases.
15. Patients with known connective tissue disorders, i.e. Lupus
16. Previous history of pericarditis
17. Presence of a PFO/ASD or valve implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of device related serious adverse events | 30 days
Percent of patients with complete exclusion of the LAA measured with TEE | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Sadowski, M.D., Ph.D, Principal Investigator — Jagiellonian University (John Paul II) Hospital
Locations (1):
- Jagiellonian University (John Paul II) Hospital, Krakow, Poland

REFERENCES:
- [Result] Bartus K, Han FT, Bednarek J, Myc J, Kapelak B, Sadowski J, Lelakowski J, Bartus S, Yakubov SJ, Lee RJ. Percutaneous left atrial appendage suture ligation using the LARIAT device in patients with atrial fibrillation: initial clinical experience. J Am Coll Cardiol. 2013 Jul 9;62(2):108-118. doi: 10.1016/j.jacc.2012.06.046. Epub 2012 Oct 10. PMID 23062528